CLINICAL TRIAL: NCT06097949
Title: The Use of a Novel Wearable Medical Device (AcuPebble SA100) to Remotely Monitor Patients With Obstructive Sleep Apnoea (OSA) on Continuous Positive Airway Pressure Therapy (CPAP)
Brief Title: AcuPebble to Remotely Monitor Patients With OSA on CPAP Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Free Hospital NHS Foundation Trust (Other)
Collaborators: Acurable Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 311874
Record Dates: First submitted 2023-09-19; First posted 2023-10-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Sleep Apnea, Obstructive
Keywords: OSA; CPAP; Wearable technology
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: AcuPebble SA100 — This device is not being used as an interventional device but simply a monitoring tool on patients already on CPAP therapy. The device is being used within the scope of it's intended purpose as a medical device to diagnose OSA.

SUMMARY:
Obstructive sleep apnoea (OSA) is a breathing problem that happens when you sleep. It is treated by a machine called continuous positive airway pressure (CPAP) therapy.

The goal of this observational trial is to test how well a new wearable device can detect ongoing OSA in patients undergoing treatment with CPAP. The main questions it aims to answer are:

1. Does the new wearable device detect OSA in patients undergoing treatment with CPAP as well as gold standard sleep studies?
2. Does the new wearable device detect OSA in patients undergoing treatment with CPAP more accurately than the CPAP machine can itself.

Participants will be asked to wear the following two devices while using their CPAP machine for 2 nights:

1. AcuPebble SA100 (the new wearable device). This device is the size of a 2-pence coin and sits on the front of the neck and attaches via some double sided sticky tape. It is connected via bluetooth to a mobile phone application (app).
2. A multi-channel sleep study, which is the gold standard way of performing sleep studies.

Researchers will then compare how much OSA is left in participants, comparing the values from the new device, gold standard sleep study and the CPAP machine itself.

DETAILED DESCRIPTION:
Obstructive sleep apnoea (OSA) affects almost one billion people globally and can lead to numerous health consequences including ischaemic heart disease, hypertension, stroke and arrhythmias. It also has a profound impact on patient's quality of life and has a high economic burden on society. Continuous positive airway pressure (CPAP) therapy is globally accepted gold-standard treatment, virtually eliminating OSA (by normalising the apnoea-hypopnoea index (AHI)), thus improving quality of life, decreasing sleepiness and reducing medical sequelae. A high residual AHI may still be present despite adequate CPAP usage in some patients. This patient population will suffer with on-going / worsening somnolence, sleep apnoea symptoms and potentially increased cardiovascular risk, which will no doubt reduce their adherence thus increasing their residual AHI, perpetuating a viscous cycle.

Currently CPAP machines can store airflow and pressure data, displaying residual events and compliance indices. However, algorithms between devices vary and there are no standards on how to use the data, and there is mixed data surrounding residual event accuracy. A review by the American Thoracic Society concluded that while CPAP usage can be reliably determined from tracking systems, residual events (residual AHI) and mask leak data are not easy to interpret and differ depending on manufactures. Some studies have found that this is especially the case in relation to detecting hypopnoeic events. Therefore, a more accurate and simple system is needed to accurately determine usage and residual events, that is: standardised, reliable and independent of machine manufacturer. Overnight oximetry is used by some Trusts as a surrogate marker of residual events. However, studies that have validated overnight oximetry against polysomnography (gold standard) have found the specificity and sensitivity decrease with decreasing severity of disease. Therefore this is not a practical or reliable way to monitor patients remotely.

Therefore we aim to assess whether we can accurately measure the residual AHI with a simple, accurate, novel wearable device in patients undergoing CPAP therapy. This will enable us to accurately assess treatment effect and highlight patients who require more intensive / change in their therapy.

AcuPebble SA100 is a CE marked novel wearable device developed by Acurable Ltd which has already been validated as an automated diagnostic tool for OSA with a high positive (96%) and high negative (995) predictive value when compared to a gold standard sleep study. This is currently in clinical use. We intend to assess whether AcuPebble SA100 can also be used to accurately detect the residual AHI in patients with OSA on CPAP therapy.

Patients in this study will be asked to wear both AcuPebble SA100 and a gold standard multi-channel sleep study simultaneously, alongside using CPAP therapy for two consecutive nights. We will then compare the residual AHI from AcuPebble SA100 with gold standard, as well as comparing the accuracy of the CPAP machine AHI with gold standard. This will also enable us to detect whether AcuPebble SA100 is more accurate that the CPAP machine.

We will also assess the usability of AcuPebble SA100 in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with an initial diagnosis of moderate/severe OSA (AHI ≥ 15events/hr made on full polysomnography, cardiorespiratory-polygraphy or other validated home sleep study) with no evidence of hypoventilation
2. Patients who have been established on CPAP therapy for > 3months
3. Patients who are deemed compliant on CPAP therapy (average use ≥ 4 hours/night for ≥ 70% of the last 28 days)

Exclusion Criteria:

* Age <18
* Subjects not fluent in English, or who have special communication needs
* Known allergy to adhesive dressing
* Subjects with physical or mental impairments who would not be able to use the device and technology on their own
* Subjects with implantable devices
* Subjects with stridor
* Subjects unable to give consent
* Subjects on non-invasive ventilation (NIV) or bi-level positive airway pressure (BIPAP)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an existing diagnosis of obstructive sleep apnoea who have been established on continuous positive airway pressure (CPAP) therapy and are deemed compliant with therapy.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2022-10-07 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the residual AHI measured by AcuPebble SA100 | 6 months
  Our primary outcome will be to measure the residual AHI with AcuPebble SA100 and compare the accuracy of this measurement against a gold standard multi-channel sleep study. The residual AHI is a measurement that quantifies the amount of sleep disordered breathing that is still present despite treatment.

SECONDARY OUTCOMES:
Comparing the residual AHI measured by AcuPebble SA100 and the CPAP machine | 6 months
  To measure the residual AHI with AcuPebble SA100 and compare it to the measurement dervied from the continuous positive airway pressure (CPAP) machine. The residual AHI is a measurement that quantifies the amount of sleep disordered breathing that is still present despite treatment.
Accuracy of the effective AHI measured by AcuPebble SA100 | 6 months
  To measure the total night-time AHI (effective AHI) using AcuPebble SA100 and compare this measurement to a gold standard multi-channel sleep study. The residual AHI is a measurement that quantifies the amount of sleep disordered breathing that is still present despite treatment.
Measure the acceptability of AcuPebble SA100 | 6 months
  To measure how comfortable AcuPebble SA100 is to wear for people while they use their CPAP machine.

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Respiratory Department Royal Free Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data